CLINICAL TRIAL: NCT01899209
Title: Obstructed Defecation Caused by Rectal Intussusception and Rectocele:STARR Versus Laparoscopic Ventral Rectopexy
Brief Title: Surgical Treatment of Obstructed Defecation Syndrome
Acronym: PRO-REST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Dajana Cuicchi, Dr Dajana Cuicchi, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-REST
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Sensation of Inadequate Defecation; Rectal Prolapse; Rectocele
Keywords: Obstructed Defecation; Rectal rectocele; Intussusception; STARR; Ventral Rectopexy
MeSH Terms: conditions — Rectal Prolapse; Rectocele; Intussusception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): STARR
  Interventions: Procedure: STARR
- Group B (Experimental): Laparoscopic ventral Rectopexy
  Interventions: Procedure: Laparoscopic Ventral Rectopexy

INTERVENTIONS:
Procedure: STARR
  Arms: Group A
Procedure: Laparoscopic Ventral Rectopexy
  Arms: Group B

SUMMARY:
Obstructed Defecation is a profoundly disabling condition. Many different surgical procedures has been introduced to treat patients affected by this disease. The most used are STARR and ventral rectopexy. Because of the heterogenity of studies and overall the lack of comparison trials, there is no accepted standard surgical treatment.PRO-REST aimed to compare these two procedures (STARR and Ventral Rectopexy) evaluating functional and anatomical results.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Obstructed Defecation with ODS score >11
* Symptomatic rectal Intussusception and/or defecographic finding of rectocele>2 cm
* Failure of at least 6 months of medical therapy
* Exclusion of neoplasm by rectosigmoidoscopy/colonoscopy

Exclusion Criteria:

* Patients affected by complete rectal prolapse
* Patients affected by slow transit constipation
* Patients affected by anismus
* Patients affected by pelvic organ prolapse
* Patients with previous rectal or anal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Functional result | 12 months
  comparison between Obstructed Defaecation Syndrome (ODS) score before and 12 months after surgery

SECONDARY OUTCOMES:
Anatomical result | 12 months
  Comparison of clinical and radiological data before and 12 months after surgery

OTHER OUTCOMES:
Quality of life and safety | 12 months
  Comparison of Constipation-Related Quality of Life questionnaire (CRQoL) before and 12 months after surgery Comparison of morbidity and mortality rate between the two procedures

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Bologna, Bologna, Italy